CLINICAL TRIAL: NCT01558128
Title: Combined Amiodarone and Electrical Cardioversion for Postoperative Atrial Fibrillation After Cardiac Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient Recruitment
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1105011705
Record Dates: First submitted 2012-03-07; First posted 2012-03-20 (Estimated); Results first posted 2017-05-23 (Actual); Last update posted 2017-05-23 (Actual); Status verified 2017-04

CONDITIONS: Cardiac Disease
MeSH Terms: conditions — Heart Diseases | interventions — Amiodarone; Electric Countershock

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Amiodarone with cardioversion (Other): If subject converts to normal sinus rhythm following amiodarone no further intervention is taken, if subject remains in atrial fibrillation following amiodarone they are cardioverted.
  Interventions: Drug: Amiodarone; Procedure: Cardioversion

INTERVENTIONS:
Drug: Amiodarone — Bolus given 150mg IV, then IV drip 1mg per hour infused for 6 hours, 0.5mg per hour infused for 18 hours.
  Other Names: Cordarone
Procedure: Cardioversion — Cardioversion done if atrial fibrillation continues following 24 hour infusion of amiodarone. Cardioversion done following hospital protocol.

SUMMARY:
To determine the efficacy of cardioversion and amiodarone for cardiac patients who develop postoperative atrial fibrillation

DETAILED DESCRIPTION:
New-onset atrial fibrillation (AF) after cardiac surgery is a well-recognized phenomenon with significant outcome implications. Incidence after coronary artery bypass grafting (CABG) is estimated at 26-33%, while those undergoing valvular surgery bear a greater burden at 33-49%. Clinical and socioeconomic complications resulting from postoperative atrial fibrillation include an increased risk of death (10%), congestive heart failure (4%), prolonged hospital stays, and increased rate of discharge to care facilities over those who remain in sinus rhythm, (7%). Although a body of evidence exists for electrical or pharmacological cardioversion to sinus rhythm postoperatively, there is a marked paucity in the literature regarding efficacy and outcomes combining the two. More specifically, we seek to evaluate the efficacy of DC cardioversion when combined with amiodarone. Improved outcomes with multimodal cardioversion may decrease the postoperative clinical burden of atrial fibrillation on cardiac surgery patients.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who underwent CABG and/or cardiac valve surgery involving cardiopulmonary bypass and develop postoperative atrial fibrillation within 7 days after surgery

Exclusion Criteria:

* Subjects who had any form of atrial fibrillation prior to surgery
* Subjects who were on antiarrhythmic medications preoperatively, including but not limited to procainamide and amiodarone

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Kerr, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Amiodarone With Cardioversion
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Amiodarone With Cardioversion
Number analyzed (Participants) | 1
Age, Continuous [Mean (Full Range); unit: years] | 87 [87 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Subject Rhythm
Description: Measuring change from baseline cardiac rhythm.
Time Frame: Participants will be followed for the duration of their hospital stay post surgery with an expected average of 7 to 10 days and again at surgical follow up appointment up to 6 weeks.
Population: Converted to normal sinus rhythm
Measure: Count of Participants; unit: Participants
Arm/Group | Amiodarone With Cardioversion
Number analyzed (Participants) | 1
Participants | 1

ADVERSE EVENTS:
Time Frame: Six weeks
Arm/Group | Amiodarone With Cardioversion
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amiodarone With Cardioversion (N=1)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No